CLINICAL TRIAL: NCT05014074
Title: The Dreamer Girls Project: Adaptation of SISTA/SIHLE for HIV/AIDS and Substance Abuse Prevention Among Black Adolescent Girls
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000026660; 2R25MH087217-11 (NIH)
Record Dates: First submitted 2021-07-19; First posted 2021-08-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: HIV/AIDS
Keywords: Black adolescent girls
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Theater/Pilot Testing (Experimental): Participants will take part in a theater/pilot testing in order to receive adequate feedback and make substantive change in the intervention
  Interventions: Other: Theater/Pilot Testing

INTERVENTIONS:
Other: Theater/Pilot Testing — Participants will take part in a theater/pilot testing in order to receive adequate feedback and make substantive change in the intervention

SUMMARY:
The study will use focus group methodology in the formative evaluation phase. Focus group methodology provides a rich source of data and understanding of phenomena by allowing the researcher to examine the interaction among participants

DETAILED DESCRIPTION:
The study is a formative qualitative study design with the intention of using findings for the adaptation and evidence-based intervention.

Study Approach: The process of modifying an evidence-based intervention (EBI) without competing with or contradicting its core elements or internal logic is referred to as ''adaptation''. To effectively implement the intervention, this study will use the ADAPT-ITT. Drs. Wingood and DiClemente have systematically developed a framework for adapting HIV-related evidence-based interventions, known as the ''ADAPT-ITT'' model. The ADAPT-ITT model consists of 8 sequential phases that inform HIV prevention providers and researchers of a prescriptive method for adapting evidence-based interventions. ADAPT-ITT has been applied with diverse populations of adolescents and adults in domestic and international settings. Due to time restrictions on the execution of this study, the first three phases of the ADAPT-ITT will be implemented.

Phase 1: Assessment involves conducting focus groups with member of the target population. For this study, it will be Black girls between the ages of 13-18 years old. The purpose of this step is to gain input from members of the target population on the intervention before it is introduced. Before implementing the adaptation of SIHLE, it is necessary for facilitators to conduct focus groups with girls who are from the target community and age group.

Phase 2: A community advisory board will be created and will involve: leaders of organizations that serve Black adolescent girls in Paterson and Black adolescent girls whom live in Paterson and are a part of the target population. The community advisory board will aid in deciding on the appropriate intervention and modify intervention components to fit the target population. Within the ADAPT-ITT framework, the next phase must include the Decision making phase. Decision phase includes deciding on which HIV intervention to implement on the target population. This stage, the PI has selected SIHLE intervention to be conducted based on a previous needs' assessment on the community. Since there are very limited interventions for Black girls that address HIV/AIDS and drug use, adapting SIHLE to fit the needs of the girls in the community will be implemented.

Phase 3: Adaptation involves using an innovative pretesting methodology known as theater testing to adapt the EBI. Using this methodology, a subset of 5-10 Black adolescent girls from the community will be invited to a central location to respond to a demonstration of the adapted SIHLE intervention.

The purpose of this registration is for Phase 3 of the study.

ELIGIBILITY:
Inclusion Criteria

1. Identify as a Black/African American female
2. Be between the ages of 13-18 years old;
3. Consent to being a part of the study (Parent consent and youth assent if under 18 years old);
4. Live in Paterson, New Jersey at the time of the study;
5. English as their first language.

Exclusion Criteria

1. not identify as Black/African American only
2. be under the age of 13 or over the age of 18
3. no parental consent provided
4. no youth assent provided
5. does not live in Paterson
6. does not read, speak or write in English
7. is currently pregnant

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — participants that identify themselves as females
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in 30-day drug use | 30 days
  Past 30-day drug use will be measured using items from the National Survey on Drug Use and Health (Substance Abuse and Mental Health Services Administration, 2006) and Youth Risk Behavior Survey. The scale consisted of three items that assesses how often participants smoked cigarettes, drank alcohol, and smoked marijuana in the past 30 days. An example of an item is, "Estimate the number of days you used marijuana or hashish in the last 30 days." Participants responded to these items on a 7-point scale (1 = 0 days; 2 =1-2 days, 3 = 3-5 days; 4 = 6-9 days; 5 = 10-19 days; 6 = 20-29 days; 7 = All 30 days). The sum of this scale is the mean of responses on the three items, with higher scores indicating greater frequency of use.
Change in perception of drug use risk | Baseline, 30 days, 60 days
  To assess the perceived risk of using alcohol, tobacco, and marijuana, adapted questions from the Monitoring the Future study will be used. Questions such as: perceived risk of moderate daily drinking, heavy drinking, combining alcohol with marijuana, daily smoking and heavy, daily and heavy marijuana use. The choices are: 0=Can't Say/Drug Unfamiliar, 1=No risk, 2=Slight risk, 3=Moderate risk, 4=Great risk. All of the items will be summed together. Higher score indicates greater perception of risk from using alcohol and drugs
Change in perception of sexual risk | Baseline, 30 days, 60 days
  Perception of Sexual Risk was assessed using eight items that measured participants' perception of sexual risk (sample item: How much do you think people risk harming themselves physically if they have sex without a condom or dental dam?) and substance use risk (sample item: How much do people risk harming themselves physically or in other ways when they smoke marijuana once or twice a week?). Items will be summed and higher scores will indicate greater perceived risk
Change in HIV knowledge | Baseline, 30 days, 60 days
  HIV Knowledge will be assessed using eight items that measured participants' HIV knowledge (sample item: Only people who look sick can spread the HIV/AIDS virus.). Responses were recorded using True (1) or False (0). Items will be summed and higher scores indicated greater HIV knowledge
Change in sexual risk behavior | Baseline, 30 days, 60 days
  Sexual Risk Behavior: Six items will be adapted from the National Youth Risk Behavior Survey , which assess sexual behavior among high school aged adolescents. These items included: having ever had vaginal sex, how many times participants had sex in the past 3 months, number of lifetime sexual partners, age of first sexual intercourse, having sex under the influence of drugs and alcohol, and having unprotected sex without a condom. A composite score will be used where the range of score is 0 to 30, the higher the score the more perception of risk
Change in ethnic identity | Baseline, 30 days, 60 days
  Multigroup Ethnic Identity Measure (MEIM) Revised consists of six questions and will be used to measure ethnic identity. Responses using a 4-point Likert-type scale will range from Strongly disagree (1) to Strongly agree (4). Scores were totaled by summing responses, with higher scores representing greater ethnic identification (Cronbach α = .86). Responses on the original MEIM ranged from 20 to a maximum of 80.

CONTACTS AND LOCATIONS:
Overall Officials: Ijeoma Opara, PhD, Principal Investigator — Yale University
Locations (1):
- Paterson Youth Services Bureau, Paterson, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Opara I, Gabriel C, Duran-Becerra B, Bond K, Hill AV, Hussett-Richardson S, Alves C, Kershaw T. Sexual Health and Drug Use Prevention for Black Girls (The Dreamer Girls Project): Protocol for an Intervention Development. JMIR Res Protoc. 2023 Aug 9;12:e45007. doi: 10.2196/45007. PMID 37556188